CLINICAL TRIAL: NCT06120010
Title: Prevalence of Anatomical Variants of Dural Sinuses by MRV Evaluation in Sohag
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Makram Sabah, Resident-Diagnostic and interventional Radiology department, Sohag University
Other Study IDs: Soh-Med-23-10-01MS
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Anatomical Variants of Dural Sinuses by MRV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — To detect prevalence of anatomical variants of dural sinuses by MRV

SUMMARY:
The purpose of this study is to use the MRV to depict the prevalence of anatomical variants of dural venous sinuses in Sohag population, which can help to avoid potenital pitfalls in the diagnosis of dural venous sinus thrombosis, venous infarcts and venous hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Sohag by nationality and residence, male or female by sex, having normal cerebral MRV reported and consented to participate in the research work will be included in this research.

Exclusion Criteria:

* Having the diagnosis of cerebral venous sinus thrombosis, congential or acquired intracranial abnormalities, ischemic or hemorrhagic stroke, intracranial hypertension, intracranial space occuping lesion, and previous head injury or neurosurgery, also patients with absolute or relative contraindications for imaging including claustrophobia, metallic implants, pacemaker and prosthetic heart valves for MRI.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Sohag by nationality and residence, male or female by sex, having normal cerebral MRV reported and consented to participate in the research work will be included in this research.
Sampling Method: Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anatomical variants of dural sinuses in Sohag population | 8 months
  Number of anatomical variants of dural sinuses by MRV evaluation in Sohag

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Dam LF, van Walderveen MAA, Kroft LJM, Kruyt ND, Wermer MJH, van Osch MJP, Huisman MV, Klok FA. Current imaging modalities for diagnosing cerebral vein thrombosis - A critical review. Thromb Res. 2020 May;189:132-139. doi: 10.1016/j.thromres.2020.03.011. Epub 2020 Mar 19. PMID 32220779
- [Background] Leach JL, Fortuna RB, Jones BV, Gaskill-Shipley MF. Imaging of cerebral venous thrombosis: current techniques, spectrum of findings, and diagnostic pitfalls. Radiographics. 2006 Oct;26 Suppl 1:S19-41; discussion S42-3. doi: 10.1148/rg.26si055174. PMID 17050515
- [Background] Cure JK, Van Tassel P, Smith MT. Normal and variant anatomy of the dural venous sinuses. Semin Ultrasound CT MR. 1994 Dec;15(6):499-519. doi: 10.1016/s0887-2171(05)80019-8. PMID 7880564
- [Background] Tubbs RS, Bosmia AN, Shoja MM, Loukas M, Cure JK, Cohen-Gadol AA. The oblique occipital sinus: a review of anatomy and imaging characteristics. Surg Radiol Anat. 2011 Nov;33(9):747-9. doi: 10.1007/s00276-011-0831-9. Epub 2011 May 29. PMID 21626273